CLINICAL TRIAL: NCT06966752
Title: Randomized Control Trial: Nasal CPAP vs. NIPPV in Preterm Infants With Respiratory Distress Syndrome
Brief Title: Comparison of Continuous Positive Airway Pressure (CPAP) and Non-Invasive Positive Pressure Ventilation (NIPPV) in Preterm Newborns With Respiratory Distress Syndrome.
Acronym: NC3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Arunas Liubsys, Associate professor, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NC3
Record Dates: First submitted 2025-03-25; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Distress Syndrome (RDS)
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP (Active Comparator): Patients under CPAP respiratory support.
  Interventions: Other: NIPPV
- NIPPV (Experimental): Patients under Noninvasive positive pressure ventilation (NIPPV).
  Interventions: Other: CPAP

INTERVENTIONS:
Other: NIPPV — NIPPV
  * PEEP 6-8 cmH2O
  * PIP: 14-16 cmH2O
  * Tinsp: 0.3-0.5sec
    * <28 weeks GA: 0.3 - 0.4 sec
    * >28weeks GA: 0.4 - 0.5 sec
  * Rate: 20-35 breaths per minute.
  Other Names: Noninvasive positive pressure ventilation
  Arms: CPAP
Other: CPAP — CPAP pressure of 6-8 mmH2O
  Other Names: Nasal Continuous Airway Pressure; nCPAP
  Arms: NIPPV

SUMMARY:
Primary objective: to evaluate safety and efficacy of two different non-invasive respiratory support modalities in preterm neonatal patients with respiratory distress syndrome.

Secondary objective is to compare different respiratory support mode performance in different gestational age groups.

Primary endpoint is treatment failure.

With this study, the following hypotheses will be tested:

Hypothesis 1: NIPPV has a lower failure rate compared to CPAP mode. Hypothesis 2: NIPPV complication rate is non-superior compared to CPAP.

DETAILED DESCRIPTION:
Treatment failure is defined as any of the following:

* FiO2>0.6 to maintain SpO2>88%
* Respiratory acidosis (pH<7.2, pCO2>65 mmHg)
* recurrent apnea (>4 episodes/h) or apnea requiring bag and mask ventilation
* Silverman Andersen respiratory severity score (SAS score) ≥6 and does not improve by > 20% within 4-8 hours

Secondary endpoints:

* Mortality rate
* Intubation rate
* Late onset sepsis (LOS) rate
* Treatment duration
* Complication rates:

Pneumothorax rate Bronchopulmonary dysplasia (BPD) Necrotizing enterocolitis (NEC) Persisting ductus arteriosus (PDA) Intraventricular hemorrhage (IVH) Retinopathy of prematurity (ROP)

Nasal trauma:

* I° - nasal/septal redness
* II° - nasal/septal redness + indent
* III° - nasal/septal redness + indent + skin breakdown

Abdominal distension:

* Visible abdominal distension (defined by attending clinician) AND one of the following:
* Feeding intolerance (defined by clinician) OR
* >3 desaturation episodes or >20% FiO2 increase in 1 hour after feed.

With this study, the following hypotheses will be tested:

Hypothesis 1: NIPPV has a lower failure rate compared to CPAP mode. Hypothesis 2: NIPPV complication rate is non-superior compared to CPAP.

ELIGIBILITY:
Inclusion Criteria:

1. gestational age (GA) between 22+0 and 34+6 weeks (estimated on the postmenstrual date and early gestation ultrasonographic findings).
2. Need of respiratory support (deemed by a clinician).

Exclusion Criteria:

1. Major congenital anomalies
2. Cardiovascular instability
3. Consent refused or not provided

Ages: 0 Minutes to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 7 days
  Need of intubation

SECONDARY OUTCOMES:
Secondary outcomes | 44 weeks corrected gestational age
  Mortality rate
Secondary outcomes | 7 days
  Intubation rate
Secondary outcomes | 44 weeks corrected gestational age
  Late onset sepsis (LOS) rate
Secondary outcomes | 44 weeks corrected gestational age
  Treatment duration
Secondary outcomes | 44 weeks corrected gestational age
  Complication rates

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Santaros Klinikos, Vilnius, Vilnius County, Lithuania

IPD SHARING:
Plan to Share IPD: No